CLINICAL TRIAL: NCT04008121
Title: A Pilot Study to Assess the Feasibility and Safety of MB-102 in Ocular Angiography as Compared to Fluorescein Sodium
Brief Title: Feasibility and Safety of MB-102 in Ocular Angiography as Compared to Fluorescein Sodium
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MB-200-01
Record Dates: First submitted 2019-05-22; First posted 2019-07-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Retinopathy; Retinal Vein Occlusion; Diabetic Retinopathy; Macular Degeneration
Keywords: Fluorescein angiography
MeSH Terms: conditions — Retinal Diseases; Retinal Vein Occlusion; Diabetic Retinopathy; Macular Degeneration | interventions — Fluorescein; relmapirazin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Adult participants with normal or diseased eyes (Experimental): 500 mg dose of intravenous fluorescein sodium followed by ocular angiography; after a minimum of 3 days, participants will receive a single intravenous dose of MB-102 at 4 μmol/kg followed by ocular angiography
  Interventions: Combination Product: Fluorescein sodium and Zeiss FF450 fundus camera; Combination Product: MB-102 and Zeiss FF450 fundus camera; Combination Product: Fluorescein sodium and commercially available optical angiography imaging system; Combination Product: MB-102 and commercially available optical angiography imaging system

INTERVENTIONS:
Combination Product: Fluorescein sodium and Zeiss FF450 fundus camera — Fluorescein sodium administered as a bolus intravenous injection; Zeiss FF450 fundus camera used for imaging of the eye of all participants
Combination Product: MB-102 and Zeiss FF450 fundus camera — MB-102 administered 3 days after fluorescein sodium as a bolus intravenous injection; Zeiss FF450 fundus camera used for imaging of the eye of all participants
Combination Product: Fluorescein sodium and commercially available optical angiography imaging system — Following Zeiss FF450 imaging, one of two systems (Heidelberg Spectralis or Optos California or 200Tx) will be used for imaging of the eye in a subset of participants
Combination Product: MB-102 and commercially available optical angiography imaging system — Following Zeiss FF450 imaging, one of two systems (Heidelberg Spectralis or Optos California or 200Tx) will be used for imaging of the eye in a subset of participants

SUMMARY:
The objective of this study is to evaluate the safety and image quality of the investigational dye, MB-102, compared to the control dye (fluorescein sodium) in healthy and diseased eyes using fluorescent angiography for retinal vascular disease diagnosis and monitoring.

DETAILED DESCRIPTION:
This will be a single-dose study, in normal participants and in those with current retinal pathology, investigating feasibility of the investigational dye, MB-102, for use in fluorescent angiography compared to fluorescein sodium. Safety and tolerability of MB-102 will also be evaluated. Control dye fluorescein sodium will be administered intravenously a minimum of 3 days prior to MB-102 dosing. After IV administration of dyes, images will be acquired of both eyes with a Zeiss fundus camera (and for some participants additional fundus photography will be performed with clinically-approved ocular angiography imaging systems) by a trained ophthalmic photographer. Participants will return for a follow-up visit after MB-102 dosing for further physical examination, clinical laboratory tests, and reporting of any adverse events. Photographs will be examined for quality as well as the utility of the angiography in evaluating disease diagnosis and progression.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years - male or female

  1. Eligible female non-pregnant participants who are either not of child-bearing potential or willing to utilize adequate contraception during the trial
  2. Males must be willing to practice abstinence or utilize adequate contraception from MB-102 dosing day to at least 7 days post dose
* Participants willing to comply with study requirements
* Participants who have signed an informed consent form

At least 5 participants will have a current history of retinal or choroidal vascular diseases.

Exclusion Criteria:

* Women who are pregnant, lactating or planning to become pregnant during the study, or women who are of childbearing potential unwilling to utilize adequate contraception
* Participation in another interventional trial within 30 days of treatment or concurrently enrolled in any other medical research study which could impact the results of the study
* History of drug or alcohol abuse within the past year
* History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, MB-102 and fluorescein sodium or other related products (intolerance to a drug is not considered a drug allergy).
* Prior history of seizures
* Current visually significant cataracts or other ophthalmic conditions that would limit appropriate collection of fundus photographs
* Site personnel immediately associated with the study or their immediate family members
* Unable to tolerate ophthalmologic imaging
* Any characteristics which, in the opinion of the investigator, makes the participant a poor candidate for participation in the clinical trial (e.g. unstable medical condition including cardiovascular disease, or other conditions considered clinically significant or unstable by the Principal Investigator)
* Prior enrollment and dosing in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Binary assessment by the Principal Investigator of the feasibility of MB-102 imaging as compared to fluorescein dye | From the time of fluorescein sodium administration through optical angiography study completion, up to 2 weeks
  Ocular angiography will be performed using a commercially available, FDA-approved clinical Zeiss FF450 fundus camera. Images will be taken of both eyes, acquired by a trained ophthalmic photographer. In at least 2 participants, imaging will also be conducted using 2 different additional clinically-approved ocular angiography imaging systems.

SECONDARY OUTCOMES:
Number of participants with adverse events | From the time of study enrollment until the end of adverse event collection, up to 24 days
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, temporally associated with the use of a medicinal product, whether or not related to the investigational drug or the reference medication. Adverse events will be collected from the time a participant is considered enrolled (after consent is signed) through the follow-up visit. Participants who fail screening will not have AEs collected.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dorshow, PhD, Study Director — MediBeacon
Locations (1):
- University of Michigan Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No